CLINICAL TRIAL: NCT00121693
Title: Posturographic Changes Associated With Music Therapy and Fall Prevention
Brief Title: The Use of Music Therapy in the Prevention of Falls
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Principal Investigator, Frederick Carrick, PhD, FACCN, Prinicipal Investigator, Carrick Institute for Graduate Studies
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CI-01-03
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Accidental Falls; Healthy
Keywords: Fall prevention; posturography; music therapy
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Music Listening 1 (Experimental): Intervention: Listen to Music type 1
  Interventions: Behavioral: Music therapy (listening to specific music)
- Music Listening 2 (Experimental): Intervention: Listen to Music type 2
  Interventions: Behavioral: Music therapy (listening to specific music)
- Music LIstening 3 (Experimental): Intervention: Listen to Music type 3
  Interventions: Behavioral: Music therapy (listening to specific music)
- Control (No Intervention): Intervention: Listen to White noise

INTERVENTIONS:
Behavioral: Music therapy (listening to specific music) — Listening to Music
  Arms: Music LIstening 3; Music Listening 1; Music Listening 2

SUMMARY:
The purpose of this study is to determine whether listening to music will demonstrate changes in human postural stability and whether those changes might be useful in fall prevention strategies.

DETAILED DESCRIPTION:
Falls are a serious health issue and are the greatest cause of death in the elderly. The use of music therapy in fall prevention has not been reported in the literature. This investigation will provide experimental support to the assumption that music therapy may prevent falls and that certain music can affect increases in postural stability using randomly selected subjects, validated posturography and a full experimental design.

Computer dynamic posturography (CDP) tests will provide stability scores in volunteer subjects who have had no previous history of falls or vertigo. Subjects will be randomized into several different music listening groups and one control group. Examiners will be blinded as to the music listened to and the outcome measurements. Subjects will be blinded as to their posturographic measurements. The music listening groups will be given a daily specific music listening task. CDP tests will be obtained 10 minutes, 1 week and 1 month after subject's treatment. Music selection will include Mozart, Nolwenn Leroy and others suggested to change human stability.

ELIGIBILITY:
Inclusion Criteria:

* No history of previous fall(s) or dizziness

Exclusion Criteria:

* History of previous fall(s) or dizziness

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2003-12; Primary Completion 2006-09 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Pretest and posttest scores will be collected for ten treatment conditions at three post-treatment times (10 minutes, 1 week, and 1 month) | Immediate pre and post balance testing
  balance testing before and after listening to music

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, FACCN, Study Director — Carrick Institute for Graduate Studies; Elena Ogerro, PhD, Principal Investigator — Carrick Institute for Graduate Studies; Guido Pagnacco, PhD, Principal Investigator — Carrick Institute for Graduate Studies
Locations (1):
- Carrick Institute for Graduate Studies, Cape Canaveral, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrick FR, Oggero E, Pagnacco G. Posturographic changes associated with music listening. J Altern Complement Med. 2007 Jun;13(5):519-26. doi: 10.1089/acm.2007.7020. PMID 17604555